CLINICAL TRIAL: NCT01214746
Title: The Effects of Atorvastatin on the Nitric Oxide-system in Healthy Young Man
Acronym: STAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: MD Frank Holden Christensen, Department of Medical Research, Regionshospitalet Holstebro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EBP-FHC-2010-1
Record Dates: First submitted 2010-05-18; First posted 2010-10-05 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Diseases; Nephropathy
Keywords: Statin; L-NMMA; Healthy subjects; Nephrology
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Placebo — 1 tablet Unikalk 1 time pr day for 5 days
  Other Names: Unikalk
  Arms: Placebo
Drug: Atorvastatin — Zarator, 80 mg pr day for 5 days
  Other Names: Zarator
  Arms: Atorvastatin

SUMMARY:
It has been documented that statin reduce mortality and morbidity in patients with cardiovascular disease. This effect can partly be related to a reduction in cholesterol levels in blood. Nitric oxide (NO) production is reduced in several chronic diseases such as nephropathy, diabetes and hypertension. The purpose of this study is to investigate the effect of Atorvastatin treatment on the NO-system measuring renal and cardiovascular variables in healthy man.

DETAILED DESCRIPTION:
Subjects will be examined on two examination days. 4 days prior to each examination day subjects are treated with either atorvastatin or placebo. During treatment periods subject are given a standardized diet.

On the examination days subject are given L-NMMA(L-NG-monomethyl Arginine citrate), a NO inhibitor, 6 mg bolus infusion followed by continuous 4 mg/kg/hr infusion for 1 hour. Renal function, central hemodynamic and vasoactive hormones are evaluated prior, during and after L-NMMA infusion.

Renal function is measured by renal clearance of 51Cr-EDTA and urinary sodium, potassium and albumin concentration. Urinary excretion of protein from sodium channels such as the NaCl cotransporter (NCC), the Na-K-Cl cotransporter (NKCC) and the epithelial sodium channel (ENaC)will be measured to evaluate channel activity in the nephron.

Central blood pressure, pulse wave analysis, and augmentation index are measured using SphygmoCor® from Atcor.

The vasoactive hormones aldosterone, renin, angiotensin II, atrial natriuretic peptide (ANP), brain natriuretic (BNP) and endothelin is measured in plasma

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18-40 years
* Body Mass Index (BMI) 18,5-30 kg/m2

Exclusion Criteria:

* Arterial hypertension (>140 mmHg systolic and/or 90 mmHg diastolic)
* Anamnestic or clinical signs of heart, lung, lever, kidney and brain disease
* Neoplastic disease
* Alcohol abuse,
* Drug abuse
* Medical treatment except oral anticontraceptive
* Smoking
* Pregnancy or
* Abnormal blood and urine sample
* Abnormal ECG
* Blood donation within a month before examination

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Fractional excretion of sodium | 5 days treatment
  Sodium excretion measured before, during and after L-NMMA infusion

SECONDARY OUTCOMES:
Systolic blood pressure (SBP) | 5 days
Pulse wave velocity | 5 days
plasma renin concentration | 5 days
Augmentation index (AI) | 5 days
Diastolic blood pressure | 5 days
Plasma aldosterone concentration | 5 days
Plasma and urinary albumin concentration | 5 days
Urinary excretion of aquaporin-2 | 5 days
plasma atrial natriuretic peptide concentration | 5 days
Plasma brain natriuretic peptide concentration | 5 days
Urinary excretion of protein from sodium channels such as the NaCl cotransporter (NCC), the Na-K-Cl cotransporter (NKCC) and the epithelial sodium channel (ENaC) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Frank H Christensen, MD, Principal Investigator — Medicinsk Forskning
Locations (1):
- Medicinsk Forskning, Regionshospitalet Holstebro, Holstebro, Denmark